CLINICAL TRIAL: NCT03940963
Title: A Multicenter, Prospective, Randomized and Subject Blinded Comparative Study of AxoGuard® Nerve Cap and Neurectomy for the Treatment of Symptomatic Neuroma and Prevention of Recurrent End-Neuroma Pain
Brief Title: Study of AxoGuard® Nerve Cap and Neurectomy for Treatment of Symptomatic Neuroma & Prevention of Recurrent Neuroma Pain
Acronym: REPOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axogen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAP-CP-001
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Symptomatic Neuroma; Morton's Neuroma; Chronic Nerve Pain
Keywords: Peripheral Nerve Injuries; Peripheral Nervous System Disease; Foot Neuroma; Foot Pain; Nerve Foot Pain; Nervous System Diseases; Trauma - Nervous System; Wounds and Injuries; Nerve Repair; Surgical Treatment of Pain
MeSH Terms: conditions — Morton Neuroma; Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Nervous System Diseases; Trauma, Nervous System; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AxoGuard® Nerve Cap (Active Comparator): Porcine derived extracellular matrix (ECM) based Nerve Termination Device.
  Excision of symptomatic neuroma of the foot or ankle with placement of Axoguard Nerve Cap over the proximal stump of the nerve.
  Interventions: Device: AxoGuard® Nerve Cap
- Standard Neurectomy (Active Comparator): Standard surgical treatment for symptomatic neuroma of the foot or ankle entailing neuroma excision (without placement of Axoguard Nerve Cap).
  Interventions: Procedure: Standard Neurectomy

INTERVENTIONS:
Device: AxoGuard® Nerve Cap — Entubulation of the nerve stump into the AxoGuard® Nerve Cap following surgical excision of symptomatic neuroma
  Arms: AxoGuard® Nerve Cap
Procedure: Standard Neurectomy — Surgical excision of symptomatic neuroma
  Arms: Standard Neurectomy

SUMMARY:
Comparing safety, pain, user experience, healthcare economic costs, work productivity, impairment and quality of life outcomes between Axoguard® Nerve Cap and neurectomy in the treatment of symptomatic neuromas in the foot or ankle. Study consists of 86 subjects randomized between the treatment groups followed for 12 months.

ELIGIBILITY:
Inclusion Criteria (Potential Subjects must):

1. Be able and willing to provide documented informed consent prior to the conduct of any study procedures;
2. Be an adult male or non-pregnant female ≥ 18 years of age;
3. Report baseline pain scores of >65mm on a 100mm Visual Analog Scale (VAS) at screening;
4. Have a documented diagnosis of symptomatic neuroma of at least one interdigital nerve in the foot which cannot be repaired to a distal nerve end;
5. Must have the of the following:

   * Pain with at least 3 of the following characteristics: burning, sharp, shooting, electric, parasthesias, numbness, cold intolerance;
   * Symptoms in a defined neural anatomic distribution
   * History of nerve injury or suspected nerve injury

   Must have at least 1:
   * Positive response to local anesthetic injection
   * US or MRI confirmation of neuroma
6. Be candidates indicated for surgery to address a symptomatic neuroma;
7. Have sufficient healthy soft tissue available to adequately cover the Axoguard® Nerve Cap;
8. In the surgeon's opinion, be likely to achieve complete resection of the symptomatic neuroma and be able to undergo implantation with the Axoguard® Nerve Cap or complete the neurotomy procedure in the control group;
9. Be willing and able to comply with all aspects of the treatment and evaluation schedule over a 12-month duration.

Exclusion Criteria (Potential Subjects must not):

1. Have undergone surgical treatment of pain from symptomatic neuroma in the target nerve(s)on three or more occasions;
2. Have biomechanical pathology and associated pain (such as plantar fasciitis, bursitis, sesamoid bone pain, tendinitis, etc);
3. Have a life expectancy of less than 12 months;
4. Have a history of or planned radiotherapy in the area of the end-neuroma;
5. be contraindicated for soft tissue implants.; this includes but is not limited to any pathology that would limit the blood supply; compromise healing or indicate the presence of a local infection;
6. Have a history of chronic ischemic conditions of the extremity;
7. Have a diagnosis of type 1 Diabetes Mellitus; or uncontrolled Type 2 Diabetes Mellitus (at the discretion of the investigator);
8. Have a history of diabetic neuropathy;
9. Be undergoing or expected to undergo treatment with chemotherapy, radiation therapy, or other known treatment which affects the growth of neural and/or vascular system;
10. Be immunosuppressed, immunocompromised or have planned immunosuppressive therapy within 12 months following the study procedure;
11. Have a History of congenital neuropathy or compressive neuropathy affecting the target limb;
12. Have a history of prior surgical management of more proximal compressive neuropathies or spinal conditions (e.g. spinal stenosis) not related to the symptomatic neuroma that affect the target limb;
13. Currently use or likely need to use medication during the study known to impact nerve regeneration or to cause peripheral neuropathy;
14. Be pregnant or plan to become pregnant during the duration of the study;
15. Be or have been enrolled in another interventional study within 30 days prior to consenting;
16. Have a known allergy to anesthetic agents;
17. Have a known sensitivity to porcine derived materials; or
18. Be, in the opinion of the Investigator, unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - New Hope Podiatry Group, Los Angeles, California
  - Anastasia Medical Group, Saint Augustine, Florida
  - EHI Clinical Research, Roswell, Georgia
  - Gateway Clinical Trials, O'Fallon, Illinois
  - OrthoIllinois, Rockford, Illinois
  - Foot and Ankle Center of Illinois, Springfield, Illinois
  - The Ohio State University, Columbus, Ohio
  - Austin Foot and Ankle Specialists, Austin, Texas
  - Complete Foot and Ankle Care of North Texas, Denton, Texas
  - JPS Health Network, Fort Worth, Texas
  - Foot & Ankle Institute, St. George, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AxoGuard® Nerve Cap: Excision of symptomatic neuroma of the foot or ankle with placement of Axoguard Nerve Cap over the proximal stump of the nerve.
Period: Overall Study
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Started | 41 | 45
Completed | 30 | 35
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population, participants that completed at least one post-baseline assessment of efficacy. Analysis was based on the treatment as received.
Groups:
- Total: Total of all reporting groups
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (11.1) | 58.7 (12.8) | 57.3 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 34 | 63
  Male | 12 | 9 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) For Pain Score at 12 Post-operative Months in Comparative Phase Subjects
Description: The Visual Analog Scale (VAS) For Pain is a patient reported outcomes scale whereby the patient indicates his/her current pain level by making a mark on a continuous horizontal 10-centimeter (100 millimeter) line. The distance from the 0 millimeter to the patient's mark corresponds to the amount of pain the participant is currently experiencing. VAS for Pain data are recorded as the number of millimeters from the left of the line to the patients mark across the range of 0-100 millimeters, with 0 millimeter representing "no pain" and 100 millimeters representing "the worst pain imaginable".
Time Frame: 12 months
Population: Intent-to-treat (ITT) population, including all participants who were randomized, received the study device or underwent neurectomy, and completed at least one post-baseline assessment of efficacy. Analysis is based on treatment as randomized.
Measure: Mean (95% Confidence Interval); unit: Millimeters (mm)
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 30 | 35
Millimeters (mm) | -86.62 [-95.21 to -78.03] | -72.67 [-81.02 to -64.32]
Statistical Analysis 1: Comparison: AxoGuard® Nerve Cap vs Standard Neurectomy; Test type: Non-Inferiority — The visual analog scale (VAS, 0-100 scale) pain score change from baseline value to 12 months was tested for non-inferiority of neurectomy with Axoguard Nerve Cap to standard neurectomy alone using closed testing procedures; p = 0.011, t-test, 2 sided — The threshold for statistical significance was p = 0.05

2. Primary Outcome: The Rate of Procedure- or Device-related Serious Adverse Events (SAEs) Through 3 Months
Description: The primary safety endpoint will compare the rate of SAEs related to the procedure or device between treatment groups. The rate of serious adverse events for a given timepoint is given as the number of participants with one or more events up to that timepoint out of the population at risk.
Time Frame: 3 months
Population: This is the safety population (SP) which includes all participants who had the study device inserted or underwent neurectomy. Analysis is based on treatment as received.
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 1 | 0

3. Primary Outcome: The Rate of Procedure- or Device-related Adverse Events (AEs) or Unanticipated Adverse Device Effects (UADEs) Through 3 Months
Description: The primary safety endpoint will compare the rate of procedure- or device-related AEs or UADEs between treatment groups. The rate of events or effects for a given timepoint is given as the number of participants with one or more events up to that timepoint out of the population at risk.
Time Frame: 3 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 4 | 4

4. Secondary Outcome: The Change From Baseline of Patient Reported Outcome Measurement Information System (PROMIS®) Pain Behavior Scale Score at Month 12
Description: The Patient Reported Outcome Measurement Information System (PROMIS®) - Pain Related Measures is a set of person-centered measures that evaluates and monitors a patient's physical health and pain. The PROMIS - pain related measures include domains evaluating fatigue, pain intensity, paint interference, sleep Disturbance, and Pain Behavior. Short forms containing fixed sets of 4-10 items or questions are included for each domain. All PROMIS scores are presented as T-scores where the T-score is the standardized score with a mean of 50 (range 20-80) and a standard deviation of 10. Higher scores indicate more of the concept being measures where sometimes the concept is desirable (e.g., physical function) and sometimes this it is undesirable (e.g., fatigue). PROMIS instruments are scored using item-level calibrations based on response patterns by HealthMeasures Scoring Service.
Time Frame: 12 months
Population: Modified intent-to-treat (mITT) population, participants that completed at least one post-baseline assessment of efficacy. Analysis is based on the treatment as received.
Measure: Mean (Inter-Quartile Range); unit: Pain Behavior Scale Score
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 30 | 35
Pain Behavior Scale Score | -19.0 [-27.2 to -14.5] | -17.1 [-28.2 to -4.6]
Statistical Analysis 1: Comparison: AxoGuard® Nerve Cap vs Standard Neurectomy; Test type: Equivalence — A predefined equivalence margin was not considered; p = 0.485, t-test, 2 sided — The threshold for statistical significance was p = 0.05

5. Secondary Outcome: Change in Foot Health Status Questionnaire (FHSQ) General Foot Health Scale at 12 Post-operative Months Compared to Baseline.
Description: The Foot Health Status Questionnaire (FHSQ) measures foot health related to quality of life based on responsiveness in overall foot health status in 4 subscale areas (foot function, foot health, footwear and foot pain). The FHSQ is comprised of 13 questions. The questionnaire is self-administered. Subscale ratings are summed and the FHSQ score is reported as 0 (poorest state of foot health) to 100 (optimal foot health) with higher scores reflecting better foot health and quality of life.
Time Frame: 12 months
Population: as for outcome 4
Measure: Mean (Inter-Quartile Range); unit: FHSQ Score
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 30 | 35
FHSQ Score | 36.7 [25.0 to 50.0] | 27.1 [0.0 to 50.0]
Statistical Analysis 1: Comparison: AxoGuard® Nerve Cap vs Standard Neurectomy; Test type: Equivalence — A predefined equivalence margin was not considered; p = 0.259, t-test, 2 sided — The threshold for statistical significance was p = 0.05

6. Secondary Outcome: As-Prescribed Opioid Medication
Description: Change from pre-operative baseline in quantity of pain medication prescribed via morphine milligram equivalent (MME) at 12 months Opioid pain medications prescribed were converted to morphine milligram equivalent (MME) where such conversions are available to summarize pain medications by quantity of use.
Time Frame: 12 Months
Population: as for outcome 4
Measure: Mean (Full Range); unit: Morphine Milligram Equivalent
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 30 | 35
Morphine Milligram Equivalent | -0.89 [-33 to 5] | 2.36 [-20 to 50]
Statistical Analysis 1: Comparison: AxoGuard® Nerve Cap vs Standard Neurectomy; Test type: Equivalence — A predefined equivalence margin was not considered; p = 0.140, t-test, 2 sided — The threshold for statistical significance was p = 0.05

7. Secondary Outcome: As-Taken Medication
Description: Change from baseline in average daily quantity of pain medication taken via the Medication Quantification Scale (MQS) at 12 months.
  A daily pain medication log was provided to each participant to take home and complete each day and was collected at all visits.
  For opioid and non-opioid pain medications, the Medication Quantification Scale (MQS) Version III is a validated tool used to quantify the complexity and detriment of pain medication regimens. It calculates a single numeric value by combining medication detriment weights (ranging from 1.1 to 4.5) with dosage levels (scaled from 1 for subtherapeutic use to 4 for supratherapeutic use). A higher MQS score indicates greater potential medication detriment and/or dosage intensity. At 12 months, the study assessed changes from baseline in patients' average daily MQS scores.
Time Frame: 12 Months
Population: Analysis population derived from modified intent-to-treat (mITT) population participants that completed at least one post-baseline assessment of efficacy and reported medications in diary. Analysis was based on the treatment as received
Measure: Mean (Inter-Quartile Range); unit: MQS Units/Day
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 24 | 26
MQS Units/Day | -1.70 [-20 to 3] | -2.43 [-15 to 1]
Statistical Analysis 1: Comparison: AxoGuard® Nerve Cap vs Standard Neurectomy; Test type: Equivalence — A predefined equivalence margin was not considered; p = 0.544, t-test, 2 sided — The threshold for statistical significance was p = 0.05

8. Secondary Outcome: Rate of Recurrence of Symptomatic Neuroma
Description: Symptomatic neuroma recurrence was defined as:
  1. VAS pain score higher at 12 months than baseline
  2. Opioid medications (MME) higher at 12 months than baseline
  3. Participant-reported pain >1 (on scale of 0-10) at least once between 9 months and 12 months.
  Participants experiencing all three of the criteria were determined to have symptomatic neuroma recurrence.
Time Frame: 12 Months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 30 | 35
Participants | 0 | 0

9. Secondary Outcome: Total Reported Pain From Baseline to 12 Months
Description: Total pain experienced by participants over the course of study follow-up was calculated from the area under the curve (AUC) of daily pain log scores reported on a 0-10 numerical rating scale. An AUC value was calculated for each participant and normalized to the total possible AUC based on the number of log entries reported for that participant. The AUC scores are reported as a proportion of the total possible AUC (on a scale of 0-1) for a participant and difference in mean treatment group values tested by a t-test.
Time Frame: 12 Months
Population: This is the per-protocol (PP) population which includes all participants in the mITT population who have an endpoint for the analysis in question and have experienced no conditions that may confound study outcomes, such as sustaining a foot injury during study follow-up. Analysis is based on the treatment as received.
Measure: Mean (Inter-Quartile Range); unit: Proportion of Area Under Pain*Time Curve
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 36 | 37
Proportion of Area Under Pain*Time Curve | 0.104 [0.019 to 0.161] | 0.187 [0.028 to 0.233]
Statistical Analysis 1: Comparison: AxoGuard® Nerve Cap vs Standard Neurectomy; Test type: Equivalence — A predefined equivalence margin was not considered; p = 0.049, t-test, 2 sided — The threshold for statistical significance was p = 0.05

10. Secondary Outcome: The Rate of Procedure- or Device-related Serious Adverse Events (SAEs) Through 6 Months
Description: The secondary safety endpoint will compare the rate of procedure- or device-related SAEs between treatment groups. The rate of serious adverse events for a given timepoint is given as the number of participants with one or more events up to that timepoint out of the population at risk.
Time Frame: 6 Months
Population: This is the safety population (SP) which includes all participants who had the study device inserted or underwent neurectomy. Treatment assignment is based on treatment as received.
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 1 | 0

11. Secondary Outcome: The Rate of Procedure- or Device-related Adverse Events (AEs) or Unanticipated Adverse Device Effects (UADEs) Through 6 Months
Description: The secondary safety endpoint will compare the rate of procedure- or device-related AEs or UADEs between treatment groups. The rate of events or effects for a given timepoint is given as the number of participants with one or more events up to that timepoint out of the population at risk.
Time Frame: 6 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 4 | 4

12. Secondary Outcome: The Rate of Procedure- or Device-related Serious Adverse Events (SAEs) Through 9 Months
Description: as for outcome 10
Time Frame: 9 Months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 1 | 0

13. Secondary Outcome: The Rate of Procedure- or Device-related Adverse Events (AEs) or Unanticipated Adverse Device Effects (UADEs) Through 9 Months
Description: as for outcome 11
Time Frame: 9 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 4 | 4

14. Secondary Outcome: The Rate of Procedure- or Device-related Serious Adverse Events (SAEs) Through 12 Months
Description: as for outcome 10
Time Frame: 12 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 1 | 0

15. Secondary Outcome: The Rate of Procedure- or Device-related Adverse Events (AEs) or Unanticipated Adverse Device Effects (UADEs) Through 12 Months
Description: as for outcome 11
Time Frame: 12 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
Number analyzed (Participants) | 41 | 43
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | AxoGuard® Nerve Cap | Standard Neurectomy
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 6/41 | 5/43
Other Adverse Events (participants affected / at risk) | 16/41 | 16/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AxoGuard® Nerve Cap (N=41) | Standard Neurectomy (N=43)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 — Determined to be unrelated to treatment
IMPAIRED HEALING (General disorders) | 1 | 0 — Anticipated risk of a surgical procedure
APPENDICITIS (Infections and infestations) | 1 | 0 — Determined to be unrelated to treatment
COVID-19 PNEUMONIA (Infections and infestations) | 1 | 0 — Determined to be unrelated to treatment
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0 — Determined to be unrelated to treatment
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 — Determined to be unrelated to treatment
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 — Determined to be unrelated to treatment
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1 — Determined to be unrelated to treatment
NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Determined to be unrelated to treatment
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 — Determined to be unrelated to treatment
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0 — Determined to be unrelated to treatment
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Determined to be unrelated to treatment
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1 — Determined to be unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AxoGuard® Nerve Cap (N=41) | Standard Neurectomy (N=43)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 1
NODULE (General disorders) | 0 | 1
OEDEMA (General disorders) | 0 | 1
PERIPHERAL SWELLING (General disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 1
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 0 | 1
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 | 1
INTENTIONAL MEDICAL DEVICE REMOVAL BY PATIENT (Injury, poisoning and procedural complications) | 1 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 1
STRESS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BURSAL FLUID ACCUMULATION (Musculoskeletal and connective tissue disorders) | 1 | 0
METATARSALGIA (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 1
PLANTAR FASCIITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1
NERVE COMPRESSION (Nervous system disorders) | 0 | 4
NEURALGIA (Nervous system disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 1
PARAESTHESIA (Nervous system disorders) | 1 | 0
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 0 | 1
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
ESSENTIAL HYPERTENSION (Vascular disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Each study site followed their standard post-operative care instructions. Variability in surgical technique for neurectomy procedures exists across study sites. The study considered sensory nerves in the foot and ankle and may be relevant to other nerve types and anatomic locations where symptomatic neuroma treatment is similar. Recurrence of neuroma was not diagnosed in the study, and additional follow-up may identify a recurrence of neuroma in some patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of at least sixty days prior to submission for publication for sponsor to review and comment. The Sponsor may extend the embargo for an additional 60 days to allow for the filing of a patent application or taking such measures Sponsor deems appropriate to establish and preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03940963/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03940963/SAP_001.pdf